CLINICAL TRIAL: NCT03925974
Title: Phase II Study of Evaluating Efficacy, Safety and Tolerance of KN026 in HER2 Expressing Advanced Gastric/Gastroesophageal Junction Cancer
Brief Title: KN026 in Patients With HER2 Expressing Gastric/Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN026-202
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Gastric/Gastroesophageal Junction Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HER2 overexpression (Experimental): HER2 IHC 3+ or IHC2+ and ISH+
  Interventions: Drug: KN026 10 mg/kg QW; Drug: KN026 20 mg/kg Q2W; Drug: KN026 30 mg/kg Q3W
- HER2 expression (Experimental): HER2 IHC 2+ISH- or IHC 1+ and ISH+
  Interventions: Drug: KN026 10 mg/kg QW; Drug: KN026 20 mg/kg Q2W; Drug: KN026 30 mg/kg Q3W

INTERVENTIONS:
Drug: KN026 10 mg/kg QW — 10 mg/kg QW as safety run-in dosage
Drug: KN026 20 mg/kg Q2W — 20 mg/kg Q2W as target dosage
Drug: KN026 30 mg/kg Q3W — 30 mg/kg Q3W as another target dosage

SUMMARY:
This is an open-label, phase 2 study of KN026 in subjects with HER2 expressing gastric/gastroesophageal junction cancer to evaluate efficacy and safety. The subjects will receive KN026 10 mg/kg QW or 20 mg/kg Q2W or 30mg/kg Q3W until progressive disease, unacceptable toxicity or death.

DETAILED DESCRIPTION:
The study consists of two arms as HER2 overexpression arm and HER2 expression arm and both arms will receive KN026 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed inform consent form(ICF)
* Age ≥ 18 years and ≤ 75 years, male or female
* Histologically or cytologically documented advanced gastric/gastroesophageal junction cancer HER2 overexpressing: IHC 3+ or IHC 2+ & ISH+ HER2 expressing: IHC2+ & ISH- or IHC 1+ & ISH+
* Received at least one prior standard therapy
* At least one evaluable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* LVEF≥ 50% (ECHO)
* Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
* Ability to comply with treatment, procedures and pharmacokinetics (PK) sample collection and the required study follow-up procedures

Exclusion Criteria:

* Accepted any other anti-tumor drug therapies within 4 weeks before fist dose
* Accepted radiotherapy within 4 weeks before enrollment
* An anthracyclines antibiotic treatment was received exceeding 320 mg/m² or other equivalent dose antharcyclines
* Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with spinal cord compression and cancerous meningitis are not eligible
* Pregnant or nursing females；or intend pregnancy within this study period or within 6 monthes after the end of this study
* History of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
* Severe chronic and active infection, need to system antibiosis/antiviral treatment
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage
* Even with peripheral or central venous nutritional support, unintentional weight loss ≥5% within 1 month before the first medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
ORR | 1 years
  clinical response rate (ORR) as determined by investigators based on RECIST 1.1 criteria
DOR | 1 years
  clinical response time (DOR) as determined by investigators based on RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China